CLINICAL TRIAL: NCT03861663
Title: Clinical Evaluation of the Next Generation Venue Ultrasound System, Components, and Accessories - Israel
Brief Title: Venue Ultrasound Evaluation - Israel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 110.04-2016-GES-0008
Record Dates: First submitted 2018-03-01; First posted 2019-03-04 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2018-12

CONDITIONS: Ultrasound Exam in Emergency/Medical Care
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Device evaluation - feasibility
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Eligible Subjects (Other): All subjects will be enrolled into a single arm and will undergo an ultrasound exam, per the protocol.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Eligible subjects will be positioned for their ultrasound exam, which will take a similar amount of time and be performed in a similar manner as standard of care ultrasound exams at the site. The type and duration of ultrasound exam will be based on the subject's clinical condition.

SUMMARY:
The study purpose is to collect images and user feedback from the Next Generation Venue Ultrasound system, components, and accessories under clinical conditions, as required for device development and optimization.

DETAILED DESCRIPTION:
Adult patients (aged >18 years) will be enrolled that present for emergency or immediate medical care, in facilities such as the intensive care unit (ICU), US unit, and/or other departments. Subjects may or may not have a clinical indication for ultrasound scanning as part of their regular medical care and will be required to meet the inclusion criteria and none of the exclusion criteria. If a subject has a clinical indication for ultrasound exam, the routine exam will be performed with the standard equipment, and an additional exam will be performed using the investigational ultrasound device.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (aged 18 years of age or older) at the time of consent;
2. Eligible to undergo ultrasound scanning per the site standard of care (with or without a clinical indication for scanning);
3. Able and willing to provide written informed consent for participation

Exclusion Criteria:

1. Are pregnant subjects
2. Require procedures that cannot be readily completed using available investigational devices;
3. Require or are anticipated to require medical care where study participation could reasonably be expected to adversely impact patient care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-01-29 (Actual); Study Completion 2018-01-29 (Actual)

PRIMARY OUTCOMES:
Obtain Image sets using Ultrasound Venue System | Two months
  Number of representative image sets for subjects enrolled in study
Periodic user feedback | Two months
  Periodic user feedback data (Clinician User Preference Survey) from device users on device performance for quality optimization. The feedback will not be aggregated or statistically analyzed. The scale is a 1-5 Likert score (1 - Poor, 2 - Needs Improvement, 3 - As expected/Equal, 4 - Better then expected, 5 - Excellent) There is no total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No